CLINICAL TRIAL: NCT03079791
Title: Prospective Registry of Impact of Level and Quality of Immunosuppression on Onset and Pattern of Cardiac Allograft Vasculopathy Evaluated by OCT.
Brief Title: Impact of Level and Quality of Immunosuppression on Onset and Pattern of Cardiac Allograft Vasculopathy Evaluated by OCT
Acronym: IMPROVE-OCT
Status: Completed | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Steffen Massberg, Prof. Dr. med., LMU Klinikum
Other Study IDs: GE MucI001-16
Record Dates: First submitted 2016-07-27; First posted 2017-03-14 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Transplant; Failure, Heart
Keywords: OCT; cardiac allograft vasculopathy; CAV; intravascular imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to use the high resolution of optical coherence tomography to assess the prevalence of different types of cardiac allograft vasculopathy (CAV) in cardiac transplanted patients and correlate those results with the level of immunosuppression

DETAILED DESCRIPTION:
CAV is the most common reason for retransplantation at >1 year and one of the main risk factors for mortality after cardiac transplantation. For this registry, patients planned to undergo coronary angiography either as a part of routine follow-up to screen for relevant cardiac allograft vasculopathy or because of clinical suspicion of relevant cardiac allograft vasculopathy will be considered eligible.

Since the "Transplant Care Guidelines of 2010" recommend the use of intracoronary imaging during angiographic follow-up in patients after heart transplantation to recognize CAV as early as possible, OCT has become integral part of the CAV diagnostic in our center. Through its high resolution OCT (so called virtual histology) provides the earliest possible diagnosis of CAV as well as new insights into the differentiation of CAV types. We aim to correlate the findings of OCT with the level of immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Patients after cardiac transplantation undergoing planed routine angiographic examination and intracoronary imaging.
* Written informed consent

Exclusion Criteria:

* Age < 18 years old
* Hemodynamic and/or electric instability
* Chronic kidney failure with glomerular filtration rate < 30 ml/min
* Pregnant or breastfeeding women
* Incapacity of providing informed consent
* If in the investigator's opinion the patient has (a) co-morbid condition(s) that could limit the patient's ability to participate in the study or impact the scientific integrity of the study
* Any contraindication to intracoronary imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after successful cardiac transplantation at the time of coronary angiography as part of routine follow-up after cardiac transplantation or as invasive diagnostic tool in case of clinical suspicion of cardiac allograft vasculopathy and indication for intravascular imaging according to guidelines.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2023-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
CAV patterns | 2 years
  Evaluation of CAV with optical coherence tomography imaging in different follow-up timepoints according to the Heart Transplant Care guidelines

SECONDARY OUTCOMES:
Immunosuppression compliance | 2 years
  Association between pattern of CAV and the appropriateness of immunosuppression as measured regularly in routine laboratory
combined ischemic events | 2 years
  Combined incidence of death, re-transplantation, myocardial infarction, stroke and coronary revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Massberg, MD, Principal Investigator — LMU Munich
Locations (1):
- Munich University Hospital, Munich, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: Undecided